CLINICAL TRIAL: NCT05158452
Title: Development of a Genetic Counseling Patient Preference Intervention for Women at Elevated Risk for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Sweet, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-20380; NCI-2021-01883 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA248739 (NIH)
Record Dates: First submitted 2021-12-03; First posted 2021-12-15 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (focus group): Participants attend a focus group over 90-120 minutes providing feedback on GCPP intervention.
  Interventions: Procedure: Discussion

INTERVENTIONS:
Procedure: Discussion — Attend a focus group
  Other Names: Discuss

SUMMARY:
This study develops a genetic counseling patient preference intervention for women at elevated risk for breast cancer. This study aims to develop an intervention that may deliver educational videos about breast cancer, heredity, multigene tests results and polygenic risk score, provide multigene and polygenic test results, obtain information about patients' questions/ concerns about test results to use in post-genetic test counseling, and determine patient preference (e.g. telephone) for receipt of post-genetic test counseling.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Develop the Genetic Counseling Patient Preference (GCPP) intervention in collaboration with community members.

OUTLINE:

Participants attend a focus group over 90-120 minutes providing feedback on GCPP intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 35-64
* Known elevated risk for breast cancer
* The ability to speak and read English
* Provide written consent

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women at elevated risk for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Development of Genetic Counseling Patient Preference (GCPP) intervention | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Sweet, MS, LGC, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu